CLINICAL TRIAL: NCT01538485
Title: Pilot Study to Assess the Effects of Vitamin D Supplementation on the Number of Regulatory FoxP3+ T Cells in the Gastrointestinal Mucosa in Healthy Women and Men: Step 3 in the Austrian Diabetes Prevention Programme
Brief Title: Vitamin D Supplementation and Regulatory FoxP3+ T Cells in the GUT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ADPP 003: GUT
Record Dates: First submitted 2012-02-08; First posted 2012-02-24 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Immune Tolerance
Keywords: Vitamin D; regulatory T cells; GUT
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cholecalciferol (Experimental)
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — weekly dose (based on 70IU KG body weight/day)
  Other Names: Oleovit D3

SUMMARY:
In this pilot study the investigators aim to investigate the effects of vitamin D supplementation on regulatory FoxP3+ T cells in the gastrointestinal mucosa in healthy women and men.

DETAILED DESCRIPTION:
This is a monocentric, open pilot study, with the aim to evaluate the effect of vitamin d supplementation on regulatory FoxP3+ T cells in the gastrointestinal mucosa in healthy women and men.

The primary goal is to evaluate the influence of vitamin D supplementation on the regulatory FoxP3+ T cells in the gastrointestinal mucosa under controlled conditions within 2 months.

The secondary study goals are to evaluate the effect of vitamin D supplementation on peripheral induced tregs and on other important immune cells in the tissue (NK, NKT cells and LPCD) and in the blood (NK, NKT cells, Th17, Th1, Th2 cells) within 2 months.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* non smoker
* BMI: 20-30 kg/m²
* Healthy

Exclusion Criteria:

* hypercalcemia > 2,65 mmol/L
* pregnancy
* chronic diseases

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Increase of regulatory FOXP3+ T cells | 2 months
  the effects of vitamin D on regulatory FOXP3+ T cells will be measured at basal and after 2 months

SECONDARY OUTCOMES:
other immune cells in the gastrointestinal mucosa | 2 months
serum calcium level | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Pieber, Prof., Principal Investigator — Medical University of Graz
Locations (1):
- Medical university Graz, Graz, Austria